CLINICAL TRIAL: NCT01379872
Title: The Assessment of New Radiation Oncology Technologies and Treatments (ANROTAT) TROG Research Project TRP11.A
Brief Title: Assessment of New Radiation Oncology Technologies and Treatments
Acronym: ANROTAT
Status: Completed | Type: Observational
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: TRP.11A
Record Dates: First submitted 2011-06-08; First posted 2011-06-23 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2011-06

CONDITIONS: Prostate Cancer (Post Prostatectomy); Anal Cancer; Nasopharyngeal Cancer; Intermediate Risk Prostate Cancer
Keywords: Prostate; Head and Neck; Anal
MeSH Terms: conditions — Prostatic Neoplasms; Anus Neoplasms; Nasopharyngeal Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Study Protocol A - IMRT Post Prostatectomy: * Prospective TROG 08.03 (RAVES) Participants
  * Prospective Participants (NOT participating in TROG 08.03 (RAVES))
  * Retrospective TROG 08.03 (RAVES) Participants
  * Participating in dosimetric evaluation and toxicity/QoL study
  * Participating in dosimetric evaluation only
  Interventions: Other: Non-Interventional Study
- Study Protocol B - IMRT Anal Cancer: * Retrospective Patient Datasets
  * Prospective Participants (dosimetric evaluation and toxicity/QoL study)
  Interventions: Other: Non-Interventional Study
- Study Protocol C - IMRT Nasopharynx: * Retrospective Patient Datasets
  * Prospective Participants (dosimetric evaluation and toxicity/QoL study)
  * Post-Treatment Prospective Participants (toxicity/QoL and cost study)
  Interventions: Other: Non-Interventional Study
- Study Protocol D - IGRT Intact Prostate: Patients with prostate cancer
  - A sample of 30 patients from at least 10 centres that are to be treated for intermediate risk prostate cancer will be enrolled. The sample will be selected to comprise at least 10 patients that will undergo non-IGRT, 10 that will undergo IGRT with fiducials and planar imaging, and 10 that will undergo IGRT with volumetric imaging.

INTERVENTIONS:
Other: Non-Interventional Study — This is a non-interventional study
  Groups: Study Protocol A - IMRT Post Prostatectomy; Study Protocol B - IMRT Anal Cancer; Study Protocol C - IMRT Nasopharynx

SUMMARY:
The Trans Tasman Radiation Oncology Group (TROG) has been commissioned by the Department of Health and Ageing to undertake a project to assess new Radiation Oncology Technology and Treatments. This project is being undertaken in response to a recognised need for the Medicare Benefits Schedule to support appropriate new radiation oncology technologies and treatments as they become available, to ensure optimal patient care.

The first phase of the project required TROG to develop a Generic Research Framework (the Framework) capable of collecting and generating information to substantiate the safety, clinical efficacy and cost effectiveness of new technologies and treatments.

The second (and current) phase of the project requires that the Framework be piloted to assess the safety, clinical efficacy and cost effectiveness of Intensity Modulated Radiation Therapy (IMRT) and Image Guided Radiation Therapy (IGRT) in four tumour site specific regions:

A. Post Prostatectomy(IMRT) B. Anal Cancer (IMRT) C. Nasopharynx (IMRT) D. Intermediate Risk Prostate Cancer (IGRT)

The aims of the site specific components of the ANROTAT protocol are as follows:

Protocol A. Develop an approach for applying the Framework to evaluate the safety, clinical efficacy and cost-effectiveness of IMRT compared to 3DCRT in patients with prostate cancer (PP).

Protocol B. Develop an approach for applying the Framework to evaluate the safety, clinical efficacy and cost-effectiveness of IMRT compared to 3DCRT in AC.

Protocol C. Develop an approach for applying the Framework to evaluate the safety, clinical efficacy and cost-effectiveness of IMRT compared to 3DCRT in NPC.

Protocol D. Develop an approach for applying the Framework to evaluate the safety, clinical efficacy and cost-effectiveness of IGRT compared to non-IGRT in patients with intermediate risk prostate cancer.

DETAILED DESCRIPTION:
The ANROTAT study is divided into four tumour site specific studies. A decision analytic model will be constructed for each disease area/technology to estimate the safety, clinical efficacy and cost effectiveness of the new technology compared to conventional standard treatment approach. This will incorporate information from previous studies and data from a series of component studies including a dosimetric evaluation, a QoL evaluation, and an evaluation of the cost of treatment planning and delivery. The development and refinement of these models is an integral component of the planned research program. The overall protocol details the data collection activities that have been identified as feasible and useful for informing the development of a series of decision analytic models to evaluate IMRT and IGRT for the four specified cancers.

These activities involve the collection of dosimetry data, quality of life (QoL) and toxicity data, and health care resource usage data in a series of component studies. These data will be used in conjunction with evidence from the existing literature and expert opinion to inform the construction of the decision analytic models.

Data will be collected from at least 10 treatment centres for each of the site specific studies. Data will be transcribed onto CRFs from source data forms. The CRFs will be sent to TROG Cancer Research on a secure fax line.

Participant's treatment plans will be securely uploaded to the TROG Central Quality Management System (CQMS) for plan review.

The data to be collected, number of participants and tasks for participants is outlined below for each of the site specific studies. WBRC has been invited to participate in Studies A and B only, however, ethics approval is sought for the entire ANROTAT protocol so our centre has approval and the option to participate in all components of ANROTAT where required.

Study Protocol A IMRT versus 3DCRT in Post Prostatectomy:

The post prostatectomy study methodology applies the ANROTAT framework and includes a series of component studies including a dosimetric evaluation, a QoL/toxicity evaluation, and an evaluation of the cost of treatment planning and delivery. This involves the collection of data from approximately 30 patients. Data collection includes eligibility, adverse events/toxicity, QoL, patient costs, and dosimetry parameters (contouring, planning, quality assurance, treatment data). These data will be used in conjunction with evidence from the existing literature and expert opinion to inform the construction of a decision analytic model.

Centres will be asked to provide two retrospective and one prospective patient but this will have to be varied according to the availability of retrospective patients at each participating centre. Each centre will be provided with details of case selection.

Data collected directly from patients will include QoL and toxicity data as well as costs incurred by the patient as a result of their treatment.

Study Protocol B IMRT versus 3DCRT in Anal Cancer:

The anal canal study methodology applies the ANROTAT framework and includes a series of component studies including a dosimetric evaluation, a QoL/toxicity evaluation, and healthcare resource usage. This involves the collection of data from 30 patients. Data collection includes eligibility, adverse events/toxicity, QoL, patient costs, and dosimetry parameters (contouring, planning, quality assurance, treatment data). These data will be used in conjunction with evidence from the existing literature and expert opinion to inform the construction of a decision analytic model.

Participating centres will be asked to provide data on the contouring and planning of a CT data set that will be sent to each of the participating centres. Following this, each participating centre will plan 3 retrospective patient cases each. In addition to this, data will be collected from 10 prospective anal cancer patients who will be asked to complete QoL and patient cost questionnaires.

Study Protocol C IMRT versus 3DCRT in NPC:

The nasopharynx study methodology applies the ANROTAT framework and includes a series of component studies including a dosimetric evaluation, a QoL/toxicity evaluation, and healthcare resource usage. This involves the collection of data from 30 patients for the dosimetry component and 150 patients for the QoL component.

Data collection includes eligibility, adverse events/toxicity, QoL, patient costs, and dosimetry parameters (contouring, planning, quality assurance, treatment data). These data will be used in conjunction with evidence from the existing literature and expert opinion to inform the construction of a decision analytic model.

Participating centres will be asked to provide data on the contouring of a CT data set that will be sent to each of the participating centres. Following this, the dosimetry component will require centres to recruit as many prospective patients as possible to collect the above mentioned data. Due to the short time frame, if 30 prospective patients cannot be recruited in the time frame, this will be supplemented with retrospective cases. In addition to this, data will be collected from 150 nasopharynx patients who will be asked to complete QoL and patient cost questionnaires.

Study Protocol D IGRT versus non IGRT in Intermediate Risk Prostate Cancer:

The IGRT study methodology applies the ANROTAT framework and includes a series of component studies including a dosimetric evaluation, a QoL/toxicity evaluation, and healthcare resource usage. This involves the collection of data from 30 prospective patients.

Data collection includes eligibility, adverse events/toxicity, QoL, patient costs, and dosimetry parameters. These data will be used in conjunction with evidence from the existing literature and expert opinion to inform the construction of a decision analytic model.

Data collected directly from patients will include QoL and toxicity data as well as costs incurred by the patient as a result of their treatment.

ELIGIBILITY:
Study Protocol A: IMRT versus 3DCRT in Post-Prostatectomy Inclusion Criteria

All of the following must apply:

* Patient has provided written informed consent
* Prior RP for adenocarcinoma of the prostate.
* Histological confirmation of adenocarcinoma of the prostate with the Gleason score reported (RP specimen).
* Patients must have at least one of the following risk factors:
* Positive margins
* Extraprostatic extension (EPE) with or without seminal vesicle involvement (pT3a or pT3b)
* PSA nadir ≤ 1.0 ng/ml following RP
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1
* Sufficient knowledge of English and adequate cognitive function to be able to complete the QoL and other questionnaires
* 18 years or older

Exclusion Criteria

None of the following must apply:

* Previous pelvic RT or surgery ie previous rectal or bladder resection
* Concurrent or previous malignancy within 5 years prior to registration (except non-melanomatous skin cancer)
* Androgen deprivation (AD) prior to or following RP as this will affect QoL
* Evidence of nodal or distant metastases
* Clinical or imaging evidence of local recurrence
* Planned adjuvant RT to cover pelvic lymph nodes
* PSA >1.0 ng/ml
* Co-morbidities that would interfere with the completion of treatment
* Concurrent cytotoxic medication
* Hip prosthesis

Study Protocol B: IMRT versus 3DCRT in Anal Cancer Inclusion Criteria

All of the following must apply:

* Informed consent for prospective patients (QoL component)
* Age 18-80 years of age
* Sufficient knowledge of English and adequate cognitive function to be able to complete the QoL and other questionnaires
* Histological confirmation of squamous cell carcinoma or basaloid carcinoma
* T2-4N0, TanyN2 (ipsilateral groin nodes) and TanyN3 (bilateral groin nodes).
* Intention to elective irradiate all pelvic nodal groups up to L5-S1 interspace (including mesorectal, presacral, internal iliac, external iliac, ischiorectal fossa, obturator and inguinal groups).
* Planned for radical chemoradiation.

Exclusion Criteria

None of the following must apply:

* Evidence of metastatic disease
* Prior pelvic RT/ surgery (e.g. vaginal hysterectomy)
* Presence of hip prosthesis
* Acquired immunodeficiency syndrome (AIDS). HIV patients without AIDS eligible.
* Previous pelvic cancers

Study Protocol C: IMRT versus 3DCRT in Nasopharynx Inclusion Criteria

All of the following must apply:

* Informed consent for prospective patients (QoL component)
* Age >18 years
* Sufficient knowledge of English and adequate cognitive function to be able to complete the QoL and other questionnaires
* Histologically confirmed carcinoma of the nasopharynx, types WHO1-111, Stage I-IVB
* Adequate staging of local disease (MRI of primary must be performed, imaging of neck nodes with CT with contrast and/or PET-CT) and exclusion of distant metastatic disease (to be confirmed by either whole body PET-CT or a chest CT, and upper abdominal CT or ultrasound scan for patients with abnormal liver function tests or a bone scan or FDG-PET for patients with bone pain).
* Disease must be considered potentially curable by chemoradiation
* Patients must be medically fit for cisplatin chemotherapy according to local practice (adequate renal, cardiac function, no significant neurological co-morbidities)
* Performance status ECOG 0, 1 or 2.

Exclusion Criteria

* Previous head and neck RT or major surgery
* Prior chemotherapy < 6 months from study entry

Study Protocol C: IGRT versus non-IGRT in Intact Prostate Inclusion Criteria

* Patient has provided written informed consent
* Aged 18 years or older
* Sufficient knowledge of English and adequate cognitive function to be able to complete the QoL and other questionnaires
* Histological diagnosis of carcinoma of the prostate < 6 months of entry without evidence of metastatic disease to the lymph nodes, bone or lung
* Intermediate risk prostate cancer (that is, T1-2a, Gleason score ≤ 6, PSA 10.1-20.0 ng/ml; T2b-c, Gleason ≤6, PSA ≤ 20.0 ng/ml; T1-2, Gleason 7, PSA ≤ 20.0 ng/ ml)

Exclusion Criteria

* Previous therapy for carcinoma of the prostate other than biopsy or transurethral resection.
* Previous pelvic RT or surgery (eg abdomino-perineal resection)
* Hip prosthesis
* Inflammatory bowel disease
* Previous or current use of AD

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Protocol A - IMRT Post Prostatectomy: Patients with prostate cancer (post prostatectomy) Study Protocol B - IMRT Anal Cancer: Patients with anal cancer Study Protocol C - IMRT Nasopharynx: Patients with nasopharynx cancer Study Protocol D - IGRT Intact Prostate: Patients with prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Comparison of dosimetry between treatment plans prepared using IMRT/IGRT vs 3DCRT/Non IGRT as a surrogate for effectiveness and safety. | 6 Months
  Measured By:
  1. Tumour control estimated from surrogate physical dose endpoints with each of the new technologies as compared with standard therapy.
  2. The likelihood of acute or long term damage to organ/tissue and resultant likelihood of impairment of function or QoL estimated from surrogate physical dose endpoints with each of the new technologies as compared with standard therapy.
Obtain Data on the impact of disease and treatment on QoL | 6 months
  Measured by
  1. QALYs gained, and cost-per-QALY gained
  2. The likely cost increases or savings resulting from differences in acute or long term toxicity.
Compare the resource usage associated with the planning and delivery of the new technologies compared to the conventional standard approaches | 6 months
  1. The differences in time and resources required for preparation, planning, quality assurance (QA) checking and treatment for each of the new technologies as compared with standard therapy.
  2. The likely cost increases or savings associated with differences in time and resources involved in the management of patients with each of the new technologies as compared with standard therapy.
Synthesise the data obtained for objectives 1-3 together with information from previous studies and expert opinion to estimate the safety, clinical efficacy and cost-effectiveness of new technologies compared to conventional standards | 6 months
  1. QALYs gained, and cost-per-QALY gained

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Burmeister, Study Chair — Trans Tasman Radiation Oncology Group
Locations (15):
- Australia (15):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Illawarra Cancer Care Centre, Wollongong, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Radiation Oncology Queensland - Toowoomba, Toowoomba, Queensland
  - Adelaide Radiotherapy Centre, Adelaide, South Australia
  - WP Holman Clinic - Royal Hobart, Hobart, Tasmania
  - WP Holman Clinic - Launceston, Launceston, Tasmania
  - Andrew Love Cancer Care Centre, Geelong Hospital, Geelong, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Hospital, Prahran, Victoria

REFERENCES:
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au